CLINICAL TRIAL: NCT00943358
Title: Safety and Immunogenicity of Cell-culture Non-adjuvanted and MF59-adjuvanted Influenza H1N1 Vaccines in Healthy Adults
Brief Title: Safety and Immunogenicity of A/H1N1v Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Public Health England (Other Government); Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UHL10763
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Influenza
Keywords: influenza; immunogenicity; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Active Comparator): adjuvanted influenza vaccine
  Interventions: Biological: MF59 H1N1 vaccine
- Vaccine 2 (Active Comparator): non-adjuvanted vaccine
  Interventions: Biological: Plain H1N1 vaccine

INTERVENTIONS:
Biological: MF59 H1N1 vaccine — 3.75-7.5ug dose
  Arms: Vaccine
Biological: Plain H1N1 vaccine — 7.5-15ug
  Arms: Vaccine 2

SUMMARY:
The purpose of this study is to evaluate the antibody response to one and two doses of influenza A/H1N1v vaccine in healthy adults.

DETAILED DESCRIPTION:
An observer-blind, single-centre study in which 7 groups of 25-30 male and female adults ≥18-50 years of age will be randomly allocated to receive two doses of cell culture non-adjuvanted or MF59-adjuvanted influenza A/California/4/2009 (H1N1) surface antigen vaccine containing 3.75, 7.5 or 15µg haemagglutinin by intramuscular injection. A second dose of the same vaccine containing the same quantity of antigen as in the first dose will be administered 21 days later. Three additional groups will receive two doses of MF59-adjuvanted influenza A/California/4/2009 (H1N1) surface antigen vaccine containing 7.5 µg haemagglutinin by intramuscular injection on day 0 or separated by 7 or 14 days. Subjects will be observed for local and systemic reactions for 30 minutes after each immunisation and will be monitored for any reactions and other adverse events for 7 days after each immunisation.

ELIGIBILITY:
Inclusion Criteria:

1. Mentally competent adults, who have signed an informed consent form after having received a detailed explanation of the study protocol.
2. Male or female subjects 18-50 years who are either healthy or have a stable medical condition.
3. Able to understand and comply with all study procedures and to complete study diaries
4. Individuals who can be contacted throughout the study and are available for all study visits
5. Females should either be using secure contraceptive precautions including:

   * the oral contraceptive pill
   * condom/barrier contraception
   * partner has had a vasectomy
   * be surgically sterilised, or
   * post-menopausal (defined as at least two years since the last menstrual period)

Exclusion Criteria:

1. Any clinically significant concurrent illness or unstable medical condition including: malignant tumours, autoimmune illnesses (including rheumatoid arthritis), acute or progressive renal or hepatic pathology, chronic obstructive pulmonary disease requiring oxygen therapy, and any active neurological disorder.
2. Individuals with a history of anaphylaxis or serious reactions to vaccines; hypersensitivity to influenzal viral protein, neomycin or polymixin, or products containing mercury.
3. Persons with known immunosuppressive disease or who use systemic immunosuppressive drugs or other drugs listed in section 8 of the British National Formulary (BNF) or chloroquine, gold or penicillamine or other drugs listed in section 10.1.3 of the BNF to suppress a chronic disease process, or have received in the last 6 months radiotherapy or chemotherapy.
4. Subjects who are at high risk of developing illnesses of the immune system.
5. Individuals who are taking immunostimulant therapy or interferon
6. Individuals who have received blood products or immunoglobulins parenterally during the preceding three months.
7. Women should not be pregnant or lactating.
8. Women who refuse to use a reliable contraceptive method throughout the study
9. Known or suspected drug abuse.
10. Individuals who have received another vaccine or investigational medicinal product in the preceding 2 weeks.
11. Unable to lead an independent life either physically or mentally
12. Regularly drink more than 40 units of alcohol weekly
13. Individuals who have had acute respiratory pathology or infections requiring systemic antibiotic or antiviral therapy during the preceding 7 days (chronic antibiotic therapy for prevention of urinary tract infections is acceptable).
14. Individuals who had a temperature >38oC in the preceding 3 days.
15. Individuals who, in the opinion of the investigator, have conditions that might complicate interpretation of the study results.
16. Individuals who have had confirmed pandemic influenza H1 infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
GMT antibody rises | 42 days

SECONDARY OUTCOMES:
frequency of adverse reactions | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Iain Stephenson, FRCP, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals Leicester, Leicester, United Kingdom

REFERENCES:
- [Derived] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215